**Date:** 1 May 2018

Study Name: Comparison Of The Incidence Of Recurrent Laryngeal Injury Following The

Dissection Of The Nerve By Cranio-Caudal And Lateral Approach By Using Introperative

**Nerve Monitoring** 

**Informed Consent Form:** 

In our research titled "Comparison of the incidence of recurrent laryngeal nerve injury following

the dissection of the nerve by cranio-caudal and lateral approach by using intraoperative nerve

monitoring", two different methods will be applied while searching for the nerve that stimulates

the vocal cords of patients planned for thyroidectomy. In the classical method, the lateral

approach nerve is sought, but as the practice of endoscopic thyroidectomy develops, the approach

to the nerve has become cranio-caudal. This study is carried out to compare the possible nerve

damage of these two methods. Our research is two-centered, will start in June 2018 and will last

until December 2019, and it is planned to include approximately 200 people in our research. You

will not be charged any fees for the methods you use in this research. In case of possible

hoarseness, your follow-up and treatment will be provided by us.

Your participation in this study can provide access to information that can reduce possible nerve

damage in thyroid surgeries, and fewer patients may experience hoarseness after surgery.

You are completely free to participate in the research or not. Not participating in this research will

certainly not affect your current treatment or the service you are receiving and your relationship

with your doctor. You have the right to withdraw by giving notice at any time; In addition, if

deemed necessary, you may be excluded from the research by the researcher, provided that your

medical condition is not harmed.

If you participate in the research, you will not be charged or charged for any expenses to be made

in the study. The sample obtained from the blood taken from you for the research will be used

only for this study. Also, at the end of the research, your information will serve scientific purposes

only, without revealing your identity.

Volunteer's Name-Surname

Signature:

Address:

Phone (Fax number):